CLINICAL TRIAL: NCT04864717
Title: A Randomized Control Trial to Compare Doxycycline to Isotretinoin for the Treatment of Acneiform Eruptions in Cancer Patients on Tyrosine Kinase Inhibitors
Brief Title: Doxycycline vs Isotretinoin for Acneiform Eruptions of TKI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Kevin Pehr, Senior Investigator/Chercheur Clinicien, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-2635
Record Dates: First submitted 2020-11-18; First posted 2021-04-29 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Acneiform Eruptions; Cancer, Treatment-Related
Keywords: Isotretinoin; Doxycyline; Tyrosine Kinase Inhibitors; EGFR Gene Mutation
MeSH Terms: conditions — Acneiform Eruptions; Neoplasms, Second Primary | interventions — Doxycycline; Isotretinoin

STUDY DESIGN:
Intervention Model Description: Two arm study: one arm isotretinoin, one arm doxycycline.
Masking Description: Unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycycline (Active Comparator): Doxycycline 100mg po once daily x 6 months
  Interventions: Drug: Doxycycline 100mg po once daily x 6 months
- Isotretinoin (Active Comparator): Isotretinoin 40mg po once daily x 6 months
  Interventions: Drug: Isotretinoin 40 mg po once daily x 6 months

INTERVENTIONS:
Drug: Doxycycline 100mg po once daily x 6 months — active intervention
  Arms: Doxycycline
Drug: Isotretinoin 40 mg po once daily x 6 months — active intervention
  Arms: Isotretinoin

SUMMARY:
Tyrosine Kinase inhibitors (TKIs) have become standard of care in patients with EGFR mutations in non-small cell lung cancer and other EGFR-mutated cancers. However, TKIs are well-known to cause cutaneous adverse events, including acneiform eruptions. Moderate to severe acneiform eruptions are often associated with severe pruritus and pain. Current treatment recommendations rely on expert consensus. Moderate and severe reactions requiring systemic therapy, usually tetracycline antibiotics or isotretinoin. No randomized trial has compared the relative effectiveness of tetracyclines versus isotretinoin.

The objective of this unblinded, randomized trial is to compare tetracyclines to isotretinoin for treatment of moderate to severe acneiform eruptions in cancer patients on tyrosine kinase inhibitors. The primary aim of this clinical trial is to elucidate which systemic treatment is more effective in clearing acneiform eruptions caused by TKIs. The results of this study will add to the literature in this field and will aid in developing evidence based clinical guidelines.

DETAILED DESCRIPTION:
Background and Study Aims:

Tyrosine Kinase inhibitors (TKIs) have become standard of care in patients with EGFR mutations in non-small cell lung cancer and other EGFR-mutated cancers. However, TKIs are well-known to cause cutaneous adverse events, including acneiform eruptions. Moderate to severe acneiform eruptions are often associated with severe pruritus and pain. Current treatment recommendations rely on expert consensus. Moderate and severe reactions requiring systemic therapy, usually tetracycline antibiotics or isotretinoin. No randomized trial has compared the relative effectiveness of tetracyclines versus isotretinoin.

The objective of this unblinded, randomized trial is to compare tetracyclines to isotretinoin for treatment of moderate to severe acneiform eruptions in cancer patients on tyrosine kinase inhibitors. The primary aim of this clinical trial is to elucidate which systemic treatment is more effective in clearing acneiform eruptions caused by TKIs. The results of this study will add to the literature in this field and will aid in developing evidence based clinical guidelines. The study will be held at Jewish General Hospital, Division of Dermatology, G026, 3755 Cote Ste Catherine, Montreal (Quebec) H3T 1E2.

Who can participate? This study is open to adult patients (>18 years old) at the Jewish General Hospital who have a histologically- or pathologically-confirmed cancer with a known sensitizing EGFR mutation. Participants must have started EGFR-TKI treatment, and subsequently had an acneiform eruption rated moderate or severe per the Leeds scale. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2, a life expectancy of at least 3 months. Premenopausal participants must use highly effective method of contraception. Female participants are neither pregnant nor breastfeeding

What does the study involve?

Participants who meet the inclusion criteria will be referred to dermatology by their treating oncologist. Participants will meet with dermatology to confirm their diagnosis, review the study protocol and ensure no exclusion criteria are met. If the participant agrees to participate in the trial, signed consent will be obtained and the participant will be randomly assigned to either the doxycycline or isotretinoin group. Participants will receive a prescription for their prescribed medication and will get the medication from their preferred pharmacy. Participants will continue regular follow up with their oncologists as per standard of care. Dermatologic study visits coincide with the follow up visit by the treating Oncologist. During these dermatology visits the following will take place:

1. Global assessment of response to skin therapy: The study dermatologist will grade the skin rash using a standardized grading system.
2. DLQI, a dermatology quality of life questionnaire
3. Participant reported new or worsening of symptoms and compliance to both the cancer medicine (TKI) and the study drug.
4. If participant consented to be photographed, follow up photographs will be obtained.
5. Routine blood tests to ensure no adverse events related to the study therapy will be reviewed.

No extra blood tests will be ordered for the study, but the blood tests already ordered by oncology will be reviewed to ensure that there are no adverse effects from the study medication. The total study duration is six months. At the end of six months, participants can choose to continue to be followed by dermatology and may continue treatment. If a participant withdraws from the study prior to six months, they will still have access to a dermatologist for treatment of the acneiform eruption.

What are the possible benefits and risks of participating? The investigators cannot guarantee that participants will receive any benefits from this study. However, this study will make an important contribution to the field of cancer care and clinical research by providing essential information on the effective treatment of common skin side effects of TKI treatment of cancer patients in the clinical setting.

Participants may have side effects from the drugs used in this study. Side effects can vary from mild to serious and may vary from person to person. Everyone taking part in the study will be watched carefully for any side effects.

All patients will be counselled on the usual adverse effects of the study medicines. In addition, specific counselling, and special emphasis, will be made for the following:

1. Pregnancy & breastfeeding. Both study medications are contra-indicated in pregnancy and breastfeeding. Pre-menopausal women will be required to use highly-effect birth control, and b-HCG will be checked with other blood tests.
2. Photosensitivity. Both study medications have a risk of photosensitivity. All patients will be counselled, and advised to use a CDA (Canadian Dermatology Association) approved sunscreen of ≥ SPF 50 at least twice daily
3. Esthetic procedures. Patients on isotretinoin will be counselled to avoid any full-depth esthetic procedures for the duration of taking the medication, plus 12 months.
4. Extreme physical exercise. Patients on isotretinoin will be counselled to avoid extreme physical exercise.
5. Mental health problems and suicide. Some patients, while taking, or soon after stopping, isotretinoin, have become depressed or developed other serious mental health problems. Signs of these problems include feelings of sadness, irritability, unusual tiredness, trouble concentrating, and loss of appetite, or even had thoughts about ending their own lives (suicidal thoughts), tried to end their own lives, and some people have ended their own lives. There were reports that some of these people did not appear depressed. There have been reports of patients on isotretinoin becoming aggressive or violent. Patients will be counselled on the importance of bringing any of the symptoms above to the attention of the study dermatologist should they arrive.
6. Neurologic (brain) problems. Patients will be asked to report symptoms of headaches, nausea, vomiting and visual disturbances given the association between isotretinoin use and benign intracranial hypertension, especially if also taking certain antibiotics (doxycycline or other tetracyclines).

Doxycycline may cause diarrhea, nausea, vomiting, exaggerated sunburn reactions, skin rash, low blood counts, liver problems, elevated intracranial pressure (which may cause changes in vision, nausea/vomiting or headaches). Some patients may develop an allergic reaction to the medication.

Isotretinoin may lead to an increase in cholesterol and triglyceride levels, liver problems, muscle pains elevated intracranial pressure (which may cause changes in vision, nausea/vomiting or headaches), abnormal development of a fetus for women who become pregnant on the medication, eye changes (dryness, decreased night vision), joint pains, pancreatitis (in patients with high blood triglyceride levels). Rarely, patients can develop a severe allergic reaction to the medication. Isotretinoin may also cause depression.

Participants will be closely monitored, including with regular bloodwork to ensure that they do not have any serious side effects to the study medications. At each visit, the study dermatologist will ask about any new symptoms that may suggest an adverse reaction to the medication. If a severe side effect develops, the study medication will be stopped and participants will be closely monitored.

Where is the study run from? The study will take place at the Jewish General Hospital in Montreal QC, Canada.

When is the study starting and how long is it expected to run for? The aim is to start the study as soon as ethics approval is obtained. The estimated start and stop dates of the trial are 01/06/2021 to 01/06/2022. The total study duration for each participant is 6 months.

Who is funding the study? There is no funding for the study.

Who is the main contact? The main contact of the study is the principal investigator. Dr. Kevin Pehr. Jewish General Hospital Senior Investigator/Chercheur Clinicien, Lady Davis Institute Associate Professor Dermatology McGill University Chief Multidisciplinary Cutaneous Lymphoma Clinic 2727B rue St Patrick Montréal (Québec) H3K 0A8 Canada (o) 514-935-1051; (c) 514-880-5122; (fax) 514-932-3793 email: kevin.pehr@mcgill.ca

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 years of age, able to understand the study procedures, and agrees to participate in the study by providing written informed consent
2. Participant has histologically- or pathologically-confirmed cancer with a known sensitizing EGFR mutation.
3. Participants must have started EGFR-TKI treatment, and subsequently had an acneiform eruption rated moderate or severe per the Leeds scale.
4. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
5. Participant has a life expectancy of at least 3 months.
6. Premenopausal participants must use highly effective method of contraception. Female participants are neither pregnant nor breastfeeding

Exclusion Criteria:

1. Absolute contraindications: pregnancy, breastfeeding, drug allergy
2. Relative contraindications:

   1. moderate to severe hypercholesterolemia (total cholesterol >7.8 mmol/L)
   2. hypertriglyceridemia (TG >2.55 mmol/L)
   3. significant hepatic dysfunction (AST > 55IU/L, ALT > 94 IU/L)
   4. suicidal ideation, pseudotumor cerebri
   5. refractory nausea or vomiting
   6. GI pathology that would prevent absorption of oral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative improvement in acneiform eruptions in cancer patients on tyrosine kinase inhibitors as defined by a change in Leeds Revised Acne Grading Scale. | 6 months
  Change in Leeds revised acne grading scale score between the baseline visit and six months or end of treatment with tyrosine kinase inhibitor, whichever is sooner. Leeds revised acne score ranges from 1 to 28, with higher being worse. Mild defined as 3-8, moderate defined as 11-20 and severe defined as 21-28.

SECONDARY OUTCOMES:
Quantitative change on patient's quality of life with treatment of the acneiform eruption as measured by the dermatology life quality index scale. | 6 months
  Patients' perception of the severity of the eruption, and its impact on their lives, before, during and after therapy using the dermatology life quality index scale, range 0-40, with higher being worse
Response of malignancy to cancer therapy using RECIST v1.1 guidelines | 6 months
  To assess response of the primary malignancy to tyrosine kinase inhibitor therapy while on the study medication using the oncology standard of care RECIST v1.1 guidelines: Complete response (CR), Partial response (PR), Stable disease (SD), Progressive disease (PD)
Adverse events from the study medications as defined using the CTCAE version 5.0 guidelines | 6 months
  To assess adverse events from combined therapy study medication and TKI using the National Institute of Health CTCAE version 5.0 guidelines. Link: https://ctep.cancer.gov/protocoldevelopment/electronic_applications/docs/ctcae_v5_quick_reference_8.5x11.pdf

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agnew T, Furber G, Leach M, Segal L. A Comprehensive Critique and Review of Published Measures of Acne Severity. J Clin Aesthet Dermatol. 2016 Jul;9(7):40-52. Epub 2016 Jul 1. PMID 27672410
- [Background] Gutzmer R, Werfel T, Mao R, Kapp A, Elsner J. Successful treatment with oral isotretinoin of acneiform skin lesions associated with cetuximab therapy. Br J Dermatol. 2005 Oct;153(4):849-51. doi: 10.1111/j.1365-2133.2005.06835.x. No abstract available. PMID 16181478
- [Background] Andrews ED, Garg N, Patel AB. A retrospective chart review on oral retinoids as a treatment for epidermal growth factor receptor inhibitor- and mitogen-activated protein kinase kinase inhibitor-induced acneiform eruptions. J Am Acad Dermatol. 2020 Apr;82(4):998-1000. doi: 10.1016/j.jaad.2019.10.003. Epub 2019 Oct 8. No abstract available. PMID 31604105
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Scope A, Agero AL, Dusza SW, Myskowski PL, Lieb JA, Saltz L, Kemeny NE, Halpern AC. Randomized double-blind trial of prophylactic oral minocycline and topical tazarotene for cetuximab-associated acne-like eruption. J Clin Oncol. 2007 Dec 1;25(34):5390-6. doi: 10.1200/JCO.2007.12.6987. PMID 18048820
- [Background] Gerber PA, Meller S, Eames T, Buhren BA, Schrumpf H, Hetzer S, Ehmann LM, Budach W, Bolke E, Matuschek C, Wollenberg A, Homey B. Management of EGFR-inhibitor associated rash: a retrospective study in 49 patients. Eur J Med Res. 2012 Feb 23;17(1):4. doi: 10.1186/2047-783X-17-4. PMID 22472354
- [Background] Lewis V, Finlay AY. 10 years experience of the Dermatology Life Quality Index (DLQI). J Investig Dermatol Symp Proc. 2004 Mar;9(2):169-80. doi: 10.1111/j.1087-0024.2004.09113.x. No abstract available. PMID 15083785
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Shikiar R, Bresnahan BW, Stone SP, Thompson C, Koo J, Revicki DA. Validity and reliability of patient reported outcomes used in psoriasis: results from two randomized clinical trials. Health Qual Life Outcomes. 2003 Oct 8;1:53. doi: 10.1186/1477-7525-1-53. PMID 14613569
- [Background] Annunziata MC, Ferrillo M, Cinelli E, Panariello L, Rocco D, Fabbrocini G. Retrospective Analysis of Skin Toxicity in Patients under Anti-EGFR Tyrosine Kinase Inhibitors: Our Experience in Lung Cancer. Open Access Maced J Med Sci. 2019 Mar 27;7(6):973-977. doi: 10.3889/oamjms.2019.170. eCollection 2019 Mar 30. PMID 30976343
- [Background] Lacouture ME. Mechanisms of cutaneous toxicities to EGFR inhibitors. Nat Rev Cancer. 2006 Oct;6(10):803-12. doi: 10.1038/nrc1970. PMID 16990857
- [Background] Melosky B, Leighl NB, Rothenstein J, Sangha R, Stewart D, Papp K. Management of egfr tki-induced dermatologic adverse events. Curr Oncol. 2015 Apr;22(2):123-32. doi: 10.3747/co.22.2430. PMID 25908911
- [Background] Giovannini M, Gregorc V, Belli C, Roca E, Lazzari C, Vigano MG, Serafico A, Villa E. Clinical Significance of Skin Toxicity due to EGFR-Targeted Therapies. J Oncol. 2009;2009:849051. doi: 10.1155/2009/849051. Epub 2009 Jun 22. PMID 19584908
- [Background] Melosky B. Supportive care treatments for toxicities of anti-egfr and other targeted agents. Curr Oncol. 2012 Jun;19(Suppl 1):S59-63. doi: 10.3747/co.19.1054. PMID 22787412
- [Background] Hirsh V. Managing treatment-related adverse events associated with egfr tyrosine kinase inhibitors in advanced non-small-cell lung cancer. Curr Oncol. 2011 Jun;18(3):126-38. doi: 10.3747/co.v18i3.877. PMID 21655159
- [Background] Sc O'brien, Jb Lewis & Wj Cunliffe (1998) The Leeds revised acne grading system, Journal of Dermatological Treatment, 9:4, 215-220, DOI: 10.3109/09546639809160698
- [Background] Bolognia, Jean., Jorizzo, Joseph L.Schaffer, Julie V., eds. Dermatology. [Philadelphia] :: Elsevier Saunders, 2012. Print.
- [Background] Ettinger DS, Wood DE, Aisner DL, Akerley W, Bauman J, Chirieac LR, D'Amico TA, DeCamp MM, Dilling TJ, Dobelbower M, Doebele RC, Govindan R, Gubens MA, Hennon M, Horn L, Komaki R, Lackner RP, Lanuti M, Leal TA, Leisch LJ, Lilenbaum R, Lin J, Loo BW Jr, Martins R, Otterson GA, Reckamp K, Riely GJ, Schild SE, Shapiro TA, Stevenson J, Swanson SJ, Tauer K, Yang SC, Gregory K, Hughes M. Non-Small Cell Lung Cancer, Version 5.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Apr;15(4):504-535. doi: 10.6004/jnccn.2017.0050. PMID 28404761
- [Background] DeWitt CA, Siroy AE, Stone SP. Acneiform eruptions associated with epidermal growth factor receptor-targeted chemotherapy. J Am Acad Dermatol. 2007 Mar;56(3):500-5. doi: 10.1016/j.jaad.2006.06.046. Epub 2006 Dec 12. PMID 17166623
- [Background] Bidoli P, Cortinovis DL, Colombo I, Crippa A, Cicchiello F, Villa F, Cazzaniga ME, Altomare G. Isotretinoin plus clindamycin seem highly effective against severe erlotinib-induced skin rash in advanced non-small cell lung cancer. J Thorac Oncol. 2010 Oct;5(10):1662-3. doi: 10.1097/JTO.0b013e3181ec1729. PMID 20871265
- [Background] Vezzoli P, Marzano AV, Onida F, Alessi E, Galassi B, Tomirotti M, Berti E. Cetuximab-induced acneiform eruption and the response to isotretinoin. Acta Derm Venereol. 2008;88(1):84-6. doi: 10.2340/00015555-0330. No abstract available. PMID 18176767
- [Background] Costello CM, Hill HE, Brumfiel CM, Yang YW, Swanson DL. Choosing between isotretinoin and acitretin for epidermal growth factor receptor inhibitor and small molecule tyrosine kinase inhibitor acneiform eruptions. J Am Acad Dermatol. 2021 Mar;84(3):840-841. doi: 10.1016/j.jaad.2020.09.090. Epub 2020 Oct 8. No abstract available. PMID 33039483
- [Background] Landis MN. Optimizing Isotretinoin Treatment of Acne: Update on Current Recommendations for Monitoring, Dosing, Safety, Adverse Effects, Compliance, and Outcomes. Am J Clin Dermatol. 2020 Jun;21(3):411-419. doi: 10.1007/s40257-020-00508-0. PMID 32107726
- [Background] Wolverton, S., 2020. Comprehensive Dermatologic Drug Therapy. 4th ed. Elsevier, pp.Chapters 9, 22. In.
- [Background] Lacouture ME, Sibaud V, Gerber PA, van den Hurk C, Fernandez-Penas P, Santini D, Jahn F, Jordan K; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Prevention and management of dermatological toxicities related to anticancer agents: ESMO Clinical Practice Guidelines☆. Ann Oncol. 2021 Feb;32(2):157-170. doi: 10.1016/j.annonc.2020.11.005. Epub 2020 Nov 25. No abstract available. PMID 33248228
- [Background] Lacouture ME, Anadkat MJ, Bensadoun RJ, Bryce J, Chan A, Epstein JB, Eaby-Sandy B, Murphy BA; MASCC Skin Toxicity Study Group. Clinical practice guidelines for the prevention and treatment of EGFR inhibitor-associated dermatologic toxicities. Support Care Cancer. 2011 Aug;19(8):1079-95. doi: 10.1007/s00520-011-1197-6. Epub 2011 Jun 1. PMID 21630130
- [Background] Cury-Martins J, Eris APM, Abdalla CMZ, Silva GB, Moura VPT, Sanches JA. Management of dermatologic adverse events from cancer therapies: recommendations of an expert panel. An Bras Dermatol. 2020 Mar-Apr;95(2):221-237. doi: 10.1016/j.abd.2020.01.001. Epub 2020 Feb 15. PMID 32165025
- [Background] Chiang HC, Anadkat MJ. Isotretinoin for high-grade or refractory epidermal growth factor receptor inhibitor-related acneiform papulopustular eruptions. J Am Acad Dermatol. 2013 Oct;69(4):657-8. doi: 10.1016/j.jaad.2013.05.032. No abstract available. PMID 24034378
- [Background] Vickers AJ, Altman DG. Statistics notes: Analysing controlled trials with baseline and follow up measurements. BMJ. 2001 Nov 10;323(7321):1123-4. doi: 10.1136/bmj.323.7321.1123. No abstract available. PMID 11701584
- [Background] O'Connell NS, Dai L, Jiang Y, Speiser JL, Ward R, Wei W, Carroll R, Gebregziabher M. Methods for Analysis of Pre-Post Data in Clinical Research: A Comparison of Five Common Methods. J Biom Biostat. 2017 Feb 24;8(1):1-8. doi: 10.4172/2155-6180.1000334. PMID 30555734
- See also: Related Info — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm